CLINICAL TRIAL: NCT02593474
Title: Medication-Assisted Treatment for Youth With Substance Use Disorders
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Elizabeth Evans, Research Psychiatrist, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #7146; U54DA037842 (NIH)
Record Dates: First submitted 2015-10-19; First posted 2015-11-02 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Opioid Use Disorder; Opioid Dependence
Keywords: Adolescent; Youth
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Naltrexone; vivitrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Detoxification / induction (Other): The detoxification / induction procedure consists of a single day of buprenorphine followed by a washout day and 4 days of ascending oral naltrexone doses. Followed on day 8 by Vivitrol injection. Participants then receive a second injection 4 weeks after the first.
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Naltrexone — Outpatient detoxification and induction onto long-acting naltrexone followed by an additional second injection of long-acting naltrexone and and additional third if desired.
  Other Names: Long acting naltrexone; Vivitrol

SUMMARY:
The purpose of this open-label pilot study is to determine the tolerability and applicability of outpatient long-acting injectable naltrexone (Vivitrol) treatment in individuals age 16-25 ("older youth") with opioid use disorder. Outpatient treatment will consist of a 7-day outpatient detoxification / naltrexone induction procedure followed by 8-weeks of treatment with Vivitrol.

DETAILED DESCRIPTION:
The rates of opioid use in youth are rising. Long-acting injectable naltrexone (Vivitrol), a medication that blocks the effects of opioid drugs, has been shown to be effective for treatment of opioid dependence in adults. Vivitrol is an important option for individuals not wanting agonist treatment (e.g. buprenorphine, methadone). Vivitrol may be particularly appealing to youth who have difficulty reaching their opioid use goals with daily oral medications as it is a monthly injection and therefore eliminates the problem of daily medication non-adherence. Vivitrol may also be appealing to families as it reduces conflicts around issues of adherence and thus supports positive parenting. Whereas Vivitrol has been used clinically in minors, it has not been studied in a prospective outpatient trial. Starting naltrexone, however, can be challenging in opioid-dependent individuals because detoxification is required prior to treatment with this medication.There are no standard outpatient detoxification protocols for opioid-dependent youth. Therefore, more studies are needed to support broader and approved use of Vivitrol in this population.

The purpose of this open-label pilot study is to determine the tolerability and applicability of outpatient long-acting injectable naltrexone (Vivitrol) treatment in individuals age 16-25 ("older youth") with opioid use disorder. We aim to have 16 older youth complete this trial. Participants will undergo an outpatient detoxification / induction procedure that has been honed over the past 13 years of work with this medication by others in our Division and is currently being used safely in opioid-dependent adults in an ongoing clinical trial. The detoxification / induction procedure consists of a single day of buprenorphine followed by a washout day and 4 days of ascending oral naltrexone doses prior to administering a dose of injectable naltrexone, typically at Day 8. Participants will then receive an additional Vivitrol injection 4 weeks after the first; they will also receive weekly medication management therapy with a research psychiatrist. Following the 9 week trial, participants and are eligible for an additional third injection followed by up to 4 weeks of therapy while proper follow-up treatment is arranged.

Primary Aim: To determine the tolerability and applicability of outpatient Vivitrol treatment in individuals aged 16-25 ("older youth") with opioid use disorder as determined by retention in treatment across the study. Outpatient treatment will consist of a 7-day detoxification / naltrexone induction procedure followed by 8-weeks of treatment with Vivitrol.

Secondary Aim 1:To determine the tolerability of 7-day outpatient detoxification / naltrexone induction for older youth as assessed by retention through first administration of Vivitrol.

Secondary Aim 2:To determine the tolerability of initial (4-week) treatment with Vivitrol as assessed by receipt of the second Vivitrol injection at week 4.

Secondary Aim 3:To determine the safety and tolerability of Vivitrol treatment as assessed with measures of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Males or females 16-25 years of age
* If adult participant (>18 y/o), capacity to provide informed consent
* If minor participants (<18 y/o), capacity to assent
* If minor participants (<18 y/o), a legal guardian available to give informed consent and accompany minor participant to all appointments or formally designate another responsible adult to accompany the minor participant to the appointments subsequent to the initial visit.
* DSM-5 criteria for opioid use disorder as a primary diagnosis
* Psychiatrically stable
* Physically healthy
* Voluntarily seeking outpatient opioid antagonist treatment
* Able to perform study procedures
* English speaking

Exclusion Criteria:

* History of allergy intolerance or hypersensitivity to the study medications
* Meets DSM-5 criteria for substance use disorder other than opioid use disorder as the primary diagnosis (except nicotine or caffeine)
* Comorbid psychiatric disorder that might interfere with or make participation hazardous, including DSM-5 diagnosis of a psychotic disorder, severe major depressive disorder, or any psychiatric disorder that may, according to the investigator's judgment, require either pharmacological or nonpharmacological intervention during the course of the study
* Pregnancy, lactation within the last 6 months, or failure to use effective contraceptive methods (condoms, diaphragm, birth control pill, IUD) in sexually active females
* Methadone maintenance treatment or regular use of illicit methadone (>30 mg per week)
* Maintenance on, or regular use of, buprenorphine or other long-acting opioid agonists
* Current suicide risk or any suicide attempts within the past year
* Unstable medical conditions or laboratory test data, which might make participation hazardous, such as acute hepatitis or ALT or AST > 3 times normal
* History of accidental drug overdose in the last three years defined as an episode of opioid-induced unconsciousness or incapacitation, whether or not medical treatment was sought or received
* Painful medical condition that requires ongoing opioid analgesia or anticipated surgery necessitating opioid medications

Ages: 16 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-04 (Actual)

PRIMARY OUTCOMES:
Retention in treatment at week 9 - the end of the study (this includes 1wk detox and 8 wks of treatment with Vivitrol) | 9 weeks

SECONDARY OUTCOMES:
Retention through first administration of Vivitrol (ie number that receive first injection) | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Evans, MD, Principal Investigator — Columbia University / New York State Psychiatric Institute
Locations (2):
- United States (2):
  - New York State Psychiatric Insitute, New York, New York
  - New York State Psychiatric Institute, New York, New York